# **5th August - 2021**

# Clinical Trials. gov PRS Protocol Registration and Results System

## "When Movement Moves" - The Health Benefits Among Individuals With Low Physical Mobility Moved by Others (WMM)

ClinicalTrials.gov ID: NCT04536779

The Ethics Committee of the Capital Region of Denmark (Human subjects protection review board)

Journal-number.: H-20010668 (Date: 13<sup>th</sup> October 2020)

# Study protocol

Title: "When Movement Moves" - The Health Benefits Among
Individuals With Low Physical Mobility Moved by Others (WMM)

## Background

Elderly and individuals with functional disabilities often face multiple personal and environmental barriers reducing their ability to engage and participate in physical and social activities [1-5]. Increasing age and level of disability correlates with lower levels of physical activity (PA), and an increased prevalence of chronic and cardiovascular diseases [6-11], which can result in premature death [12-15]. Contemporary literature indicates a dose-response relationship between PA and promotion of all health outcomes: the greatest risk reduction comes with higher intensities of PA [16], thus, PA serves as disease prevention and health maintenance [6, 17]. Moreover, the World Health Organisation encourages elderlies and disabled, regardless of age or impairments, to perform any kind of PA, as 'some is better than nothing' [18]. Additionally, a recent review indicates that less PA than the recommended can enhance health outcomes among persons with a disability [19]. Moreover, a recent study has linked various alternative forms of PA and therapy to be beneficial for health promotion and rehabilitation among individuals with cerebral palsy (CP) [20]. The literature further indicates that PA can promote cognitive function among the elderly [21] and cognitively disabled [22] on top of the well-known physiological benefits of PA. Elderly and disabled persons participating in adapted sports experience an increase to mental and social health factors, e.g., decreased feelings of loneliness, increased feelings of self-efficacy [23], autonomy and well-being [24, 25] and improvements in quality of life (QoL) [25-29]. Social support is identified as a crucial facilitator of the disabled and elderly's participation in PA [30]. Prior studies, however, have mainly focused on individuals with spinal cord injuries or elderly who can participate in (elite)sport and PA by themselves, despite a disability [24, 27, 31] or physical limitations due ageing [32]. There is a lack of literature on the frailest individuals in these groups, who are unable to participate in most kinds of PA. The few studies available have low external (i.e generalisability) validity [27, 33]. Pilot studies investigating indirect PA (defined as an activity where a person unable to partake in physical activity on their own, is joined by someone who is

able, and together partake in PA) in the disabled [34] and elderly [35-40] populations exist, however, and these report promising effects of indirect PA on all health outcomes and QoL

Despite the existence of pilot studies, little is known about the physical, mental and social health benefits of participation in indirect PA in a social context. Programmes (interventions/initiatives) providing indirect PA may motivate and promote participation if (some of) the same health benefits derived from PA can be attained through indirect PA, which may in turn result in improved QoL of the elderly and disabled. Therefore, the research project "When Movement Moves" (WMM) evaluates the pre-existing Danish programmes: Team Twin (TT) and Cycling Without Age (CWA) as both programmes make use of volunteers to assist indirect PA in disabled individuals and the elderly, respectively, using equipment designed for the purpose. The programmes ultimately share the same goal: enhancement of QoL and promotion of physical, social and mental health achieved through indirect PA in a social context [41, 42].

#### Aim

The overall hypothesis is that the activities delivered by Team Twin and Cycling Without Age increase the quality of life of the participants who are moved through others. The purpose of the trial is to investigate the physiological, mental, social health effect among individuals with low physical mobility participating in one of the two pre-existing initiatives: the Danish 'Team Twin' and Cycling Without Age. In these, the individuals with low physical mobility are moved by and together with normal functioning volunteers. Furthermore, we will investigate the importance of being a volunteer runner and pilot, relatives of and care staff for disabled athletes and the elderly.

Based on the above, this research project will answer the following research questions:

- 1. Does movement by others improves the quality of life (QOL) among individuals with low physical mobility
- 2. Does movement by others improves the physiological health among individuals with low physical mobility
- 3. Does moving individuals with low physical mobility improve health among normal functioning individuals (i.e volunteer runners and pilots)?
- 4. How does participation in the physical activity initiatives influence well-being, relations and attitudes among relatives (to the disabled individuals) and employees at nursing homes?

## Design and Methods

#### Settings

The WMM-project will be conducted in collaboration with the local departments of Team Twin (TT) and Cycling Without Age (CWA).

#### The Team Twin association

The TT association is the overall umbrella-organization for the sports and inclusion concept "Team Twin — We run Together". It was established in the year of 2014. Since then, the TT association have grown, and the association now has local departments established all over Denmark with the biggest local department located in Copenhagen with approximately 100 members [43]. The total amount of local department has grown to nine since the beginning and has over 400 members in varied age, disabled and non-disabled, women, men, adolescence and adults (for an overview of the organization chart of the Team Twin association see figure 1). The intensity, exercises (triathlete inspired), and duration can vary from club to club and according to time of the season. Handicap Athletes and voluenteers, so called runners, are expected to participate in a minimum of 8-10 training sessions during the trial period, which is a minimum of 3 months. In the period from Oktober 2020 to January 2021, two-three new local departments are expected to be established. In close cooperation between Team Twin and Institute of Public Health , Uiversity of Southern Denmark (SDU), we will seek out to recruit the recent members of the latest established local departments of TT.

The details of times and investigations will be determined in collaboration with the local associations and with regard to planned training courses and possible participation in competitions.

#### Cycling Without Age

Cycling Without Age is a worldwide association started up in Denmark, whose mission is to give the elderly "the right to wind their hair". Volunteers, so-called pilots, cycle elderly people, so called passengers, with low level of mobility in rickshaws on shorter or longer trips. The primary purpose is to give senior citizens a feeling of joy and give them the opportunity to remain an active part of the community. In Denmark, there are more than 7,000 volunteer pilots across 430 locations, typically care centers, with a total of 500 rickshaws. In 2018, a total of 14,877 registered bicycle trips were made [42].

A minimum of 6-8 bicycle trips during the intervention period, which is a minimum of 3 months, is, however, assumed to be necessary in order to be able to attribute the effect to the intervention. The

details of times and examinations will be determined in collaboration with the local care centers and any planned bicycle trips.

#### Theoretic framework for evaluation

The programme theory Illustrates the causal chain, which explains the hypothesis of how the intervention components of the Team Twin and Cycling Without Age are expected to impact the participants quality of life by participating in one of the two components (Figure 1).



Figure 1 Overall program theory for WMM-study

Quality of life is a broad concept, and there are many different definitions, all of which include dimensions of physical, social and mental health. The World Health Organization (WHO) defines quality of life as: "..an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. It is a broad ranging concept affected in a complex way by the person's physical health, psychological state, personal beliefs, social relationships and their relationship to salient features of their environment." [44] Qualilty of life will be elucidated from different angles and examined by different quantitative and qualitative methods such as through a) scientific methods in the form of physiological measurements and physical tests b) questionnaires and c) interviews and observations.

#### Study designs

The WWM-study consists of different parts and each part has its own approach, methods and measures, which will be described below. Prior to the data collection, we will pilot test our questionaries, interviewand observation guides for the potential adjustments according to the data collection methods. Further, we will conduct a minor pilot test of the laboratory protocol with 1-2 Handiathletes affiliated in an existing local department of Team Twin. The study has been reported to the Danish National Committee on Health Research Ethics Journal-nr.: H-20010668 ().

The target groups of the WMM trial are: 1) Handiathletes (Team Twin) and Passengers (Cycling Without Age and 2) the volunteer persons called "Runners" (TT) and "pilots" (CWA), who are the persons who move the diabled, Relatives (i.e. parents and siblings of the Handiathletes and 4) Nursing Staff (e.g. NS working at a care home, disabled carer or disabled escort for elderlies). The disabilities among the Handiathletes varies but the three most common are 1) cerebral palsy, 2) muscular dystrophy and 3) non-specific inherent faulty genes. Amog the elderly, it will mainly be age-related mobility decline however, also some decrease in cognitive functioning occurs among some of the participants.

#### Sub-study 1. Team Twin

**Study design**: Self-controlled before and after study. We do not consider it practically possible to carry out a study with a control group due to the relatively modest number of new members in the association.

**Target group**: Handiathletes (n=25) and runners (n=25). For the explorative study, inteviews will be conducted with Handiathletes (n=4-6) and runners (n=4-6). Also, relatives will be included in focus group interviews (n=4-7).

**Methods**: Physiological measurements and questionnaire with three measurement points. Twice before the start of the training course and once immediately after the end of the training course. This means that the individual participant acts as his or her own control. This sub study consist of two parts 1) a pre-post short-term effect evaluation; and 2) an explorative study guided by the program theory, in which examine how, why and what has an impact on mental and social health.

**Study period**: The baseline measure for this substudy is medio February 2021 (before the training season), and follow-up measurements will be conducted four months later in ultimo June.

**Primary outcomes**: Quality of Life for Handiathletes and secondarily the physiological effects.

#### Measurements:

Selfreported Questionaire (Handi Athletes, Runners and relatives): Quality of Life will be measured by questionnaire. For detailed information on the questionnaire, see the measurements section below.

Weekly text-message (SMS) (Handiathletes and Runners): registration of perceived well-being and quality of life.

Movement sensors (Handiathletes and Runners): Heart rate registration (GARMIN-watch). Runners will be informed, and trained in the use of the technology. The a GARMIN-watch will be attached to the wrist of the Handiathletes to quantify the level of physical activity during training and races throw the trial period. Further, the Garmin-watch will monitor the quality of sleep for one week in the trial period.

Clinical test (Handiathletes only): 1) Dual x-ray absorptiometry (DXA -scan) for measure change in body composition (body fat and lean mass), 2) Blood samples for measuring the metabolic change including; serum concentration of cholesterols, triglycerides, glucose, C-peptide, insulin and HbA1c, haematology, electrolytes, metabolites, liver- and renal status, endocrinology (including HCG if relevant) and markers of immune function/inflammatory, 3) Oral glucose tolerance test (OGTT) will be performed for screening the glucose level (metabolism inflammation: plasma- LDL, HDL, TG, TC, fasting insulin, C-peptide and glucose), 4) Blood volume (BV) status will be conducted to investigate the training effects on central underlying mechanisms of cardiorespiratory fitness, namely, total BV, plasma volume (PV) and haemoglobin mass (Hbmass).

*Interviews (Focusgroup and single interviews) and observations*: For detailed information on the interviews and observations, see the measurements section below.



Overview of activities taking place during the TT subproject of WMM  $\,$ 

#### Sub-study 2 – Cycling without age

**Study design**: Before and after evaluation of the Cycling Without Age activities on Quality of life using matching-adjusted indirect comparison between elderlies enrolled with the activities and elderlies not enrolled. This design is chosen, as randomization is not considered a realistic option in this real world pragmatic trial.

**Target group**: Passengers (Elderlies at nursing homes) (n=aprrox. 100 in the 'intervention group')) and piltos (n=approx. 100). In close collaboration with the association Cycling Without Age, we will recruit participants for the research project. We will strive to include older people who have not previously participated in activities with Cycling Without Age.

**Methods**: Selfreported questionnaire before and after the activities (at least two measuremnets). We will monitor whether it is possible to observe a dose-response relationship eg. Duration and distance.

**Study period**: The baseline measure for this substudy is spring 2021.

**Primary outcomes**: Quality of Life for elderlies. Secondary outcomes: mental, physical, and social health. (See program theory)

#### Measurements:

This section will explain the characteristics of the material and instruments used to conduct a quantitative investigation of the Cycling Without Age subproject.

Objective Functional and Cognitive Appraisal: A test battery will be conducted pre and post on-site at the participants' residence to evaluate a change in cognitive and physical function among nursing home residents. Cognitive function Brief Assessment of Impaired Cognition Questionnaire (BASIC-Q). A simple and newly invented tool for practitioners and healthcare professionals was selected to assess a possible change in the cognitive function level of the nursing home residents

Physical Function and Mobility: To evaluate physical performance and a possible change frompre to post, various physical tests were selected. Our test battery includes (1) the Short Physical Performance Battery, (2) the 4 m gait speed test and (3) the 6-min walking test (6MWT). The battery is performed on-site, where the nursing home resident lives, following recommended guidelines and standard procedures for each test [75,76]. All the tests are highly recommended in research and used among elderlies to detect functional capacity and sarcopenia symptoms. The chosen tests have shown great validity and reliability [77].

Muscle Strength; Muscle strength will be evaluated with (1) the chair and stand test (which is incorporated in SPPB) and (2) handgrip strength. The grip-strength measure is performed three times with a 1-min interval between each attempt. The attempt with the highest score (measured in kilograms) will count as the final.

#### Power Calculation

Based on a Danish Ph.D. project from 2019 [45], our study should include a minimum of 19 Handi Athletes, to detect a 10% increased effect in the main outcome (Quality of Life) (effect size 10%, absolute change 0.66, standard deviation 1.0, strength (beta): 0.8, alpha: 0.05). However, the WMM-study aim to recruit more than 19 Handiathletes to participate in the questionnaire (Sub study 2 and 3).



Overview of activities taking place during the CWA sub-project of WMM

#### Data collection methods

#### Questionaries

The questionaries are mainly based on validated measures (i.a. Cantril Ladder of Life Scale WHOQOL-disability modul, WHO-5 and (S)WEMWBS), further, it will be supplemented with items from other studies including EQOL[45] and SHILD[46]. "Cantrills Ladder" is used and validated in a lot of studies as a simple way to ask people to rate their current satisfaction with life - or happiness from a scale from 0-10 (where 10 is the best and most satisfying life you can have, and 0 I vice versa)[47]. Therefore, this scale is expected to a validated measure tool that can be used among many different target groups – including WMM.

New items will be developed especially related to the WMM-Study to uncover the study hypothesizes. The questionnaires will cover themes in the overall and taget group specific program theory. The questionnaire will be developed among the research group, expert group and internal colleagues who have research experience with the target group.

The questionnaire for the Runners and pilots seeks to measure the volunteers Qulaity of life and the underlying sub-themes according to Quality of Life. The questionnaire will be developed by the research group and will seek inspiration from other studies i.e the ABC-mental health study[48]. The questionnaire will cover the following themes: QOL, life satisfaction, Identity self-assessed health, Physical activity and social cohesion, welfare, voluntariness, value & importance. Also the questionaire to the relatives and the Nursing staff will cover the following some of the above menstioned themes.

#### Observations

For each of the sub study we observe 6-8 activities, where we cycle and run with the participants to get insight into how the activities proceed, the effects on mood and on how the participants interact. Insights from the participant observations are expected to feed into the subsequent interviews with the participants and give us a unique opportunity to follow up on specific elements, episodes and participant reactions in the courses. Participant observation is particularly well suited to examining social processes and concrete interactions and participant reactions in situ.

#### Interviews

To obtain the participants' descriptions of their experiences, qualitative interviews will be conducted with the disabled athletes (n = 4-6) and the runners (n = 4-6) (Team Twin) as well as with the passengers (n = 4-6) and pilots (n = 4-6) (Cycling Without Age). The interviews are conducted 4-5 weeks after the beginning of the activities using semi-structured, individual interviews, which are suitable for exploratory studies, where

the informants' experiences, perspectives, reasoning and ways of talking about the phenomenon under investigation are in focus.

Also, four focus group interviews will be conducted (n = 4-7) with relatives and caregivers. Focus group interviews are suitable for shedding light on different experiences and perspectives on a given research topic.

For all interviews, an interview guide is developed based on the research questions and adapted to the target group. Recruitment of the participants and sampling takes place in collaboration with Team Tvilling and Cycling Without Age associations. The empirical material (transcripts of interviews and field notes) is analyzed according to general principles of qualitative analysis.

#### Trial period and Organization

The project will be coordinated from 2020 to 2023 by the Center for Intervention Research at the National Institute of Public Health, SDU. The National Institute of Public Health has set up an interdisciplinary project group that has extensive experience with research into physical activity as well as mental health and quality of life, including the importance of meaningful communities. Acitivities will be carried out in close collaboration with the Team Twin and the Cycling Without Age associations. TrygFonden's Centre for Physical Activity Research (CFAS) is included as a project partner and will be responsible for the laboratory testing of people with physical disabilities.

#### Founding

The study is founded by financial support from the Bevica Foundation (2.5 mill DKK) and Helsefonden (2.5 mill DKK).

#### **Ethics Consideration**

The WMM study s will be registered in the Danish research ethics committee and data protection agency (awaiting number of registration). It will be guided and reported in accordance to the CONSORT declaration (Consolidated Standards of Reporting Trials). The trial will follow the European General Data Protection Regulation (GDPR), and the guidelines from the "Danish Council for Independent Research". Regarding the target group, the project will take their different condition in for consideration at all stages of the project.

## Statistical Analysis Plan (SAP)

Changes from pre to post in mean score of QoL, measured using Cantril's Ladder [47, 49], will be the primary statistical outcome measure. Secondary outcomes will include sleep, well-being, loneliness and autonomy, as these were identified, during our design phase, to be essential factors for the target groups. In addition, changes in the objective measures (clinical examination and physical function test) will also be conducted for each target group. For descriptive statistics and to inform participant characteristics, we plan to use paired t-tests and chi-square tests. We furthermore intend to conduct regression analyses, using a mixed method approach to compare pre and post messures. Analyses will be performed as perprotocol and after the intention-to-treat principle, which, in this case, means that potential dropouts (with incomplete data) are included in the analyses. Per-protocol participants are defined as participants who have participated in a minimum of eight TT or CWA-activities in the period from pre to post measurements. The analyses will be adjusted for sociodemographic factors such as sex, age and educational level. Data is analysed using significance levels of p=0.05 and 95% confidence intervals. Analyses will be completed by Stata Software (StataCorp LP, College Station, Texas).

# Outcomes measures and approaches Sub-study 1. Team Twin

#### Outcomes and measures in the Team Twin evaluation

| Measurement<br>(outcome) | What (operational) | How (instrument) | When<br>(timing of<br>collection) | Who in CWA<br>(Data source) |
|---|---|---|---|---|
| PRIMARY OUTCOME | | | | |
| Quality of life (QoL) | Cantril Ladder of Life Scale<br>[49] | Web- and interview-<br>based questionnaire | Baseline, follow-up | Passengers, Pilots,<br>Nursing staff |
| SECONDARY OUTCOMES | | | | |
| Autonomy | The perceived feeling of being in control over ones own life | Web-based<br>questionnaire | Baseline, follow-up | Passengers |
| Sleep | Sleep quality and sleep quantity | Web-based<br>questionnaire | Baseline, follow-up | Passengers, Pilots, |

| Measurement<br>(outcome) | What (operational) | How (instrument) | When<br>(timing of<br>collection) | Who in CWA<br>(Data source) |
|---|---|---|---|---|
| Well-being | CUA: Warwick-<br>Edinburgh Mental<br>Well- Being Scale<br>(S)WEMWBS) [50, 51] | Web-based<br>questionnaire | Baseline, follow-up | Passengers, Pilots |
| Loneliness | A perceived feeling of loneliness and lack of network and support [52, 53] | Web-based<br>questionnaire | Baseline, follow-up | Passengers, Pilots |
| EXPLORATIVE OUTCOM | ES | | | |
| Self-perceived<br>health | Subjectively perceived<br>Health [54] | Web-based questionnaire | Baseline, follow-up | Passengers, Pilots, |
| Perceived pain | Mental and physical pain/discomfort [54] | Web-based questionnaire | Baseline, follow-up | Passengers, pilots |
| Self-perceived<br>Physical performance | Subjectively perceived<br>Physical performance<br>[55] | Web-based<br>questionnaire | Baseline, follow-up | Passengers, pilots |
| Self-efficacy | General self-efficacy [56,<br>57] | Web-based<br>questionnaire | Baseline, follow-up | Passengers, pilots |
| Self-worth | Perceived feeling of<br>Acceptance [45] | Web-based<br>questionnaire | Baseline, follow-up | Passengers, pilots |
| Autonomy | The perceived feeling of being in control over ones own life | Web-based<br>questionnaire | Baseline, follow-up | Passengers, pilots |
| Social/emotional support and network | Contact and support with friends, family and others. The perceived feeling of being valued, respected and accepted by others [54] | Web-based<br>questionnaire | Baseline, follow-up | Passengers, pilots |
| UNINTENDED SIDE EFFE | CCTS | 1 | 1 | ı |
| Fatigue | The perceived feeling of fatigue related to voluntariness or programme activity | Web-based<br>questionnaire | Follow-up | Passengers, pilots |
| Anxiety | The perceived feeling of anxiety trigged by the programme activity | Web-based<br>questionnaire | Follow-up | Passengers, pilots |

| Measurement<br>(outcome) | What (operational) | How (instrument) | When<br>(timing of<br>collection) | Who in CWA<br>(Data source) |
|---|---|---|---|---|
| Injuries | Amount of injuries by participation | Web-based questionnaire | Follow-up | Passengers, pilots |
| Objective functional and | d cognitive level (only for CW) | A; Passengers) | | |
| Cognitive function | Brief Assessment of<br>Impaired Cognition<br>Questionnaire (BASIC-Q)<br>[58, 59] | Interview based case-<br>findings survey | Baseline, follow-up | Passengers |
| Physical function and mobility | Short Physical<br>Performance Battery<br>(SPPB) [60, 61] | Functional and physical test | Baseline, follow-up | Passengers |
| Muscle Strength | Grip Strength [62] | Physical test | Baseline, follow-up | Passengers |
| Gait endurance | 6-Minute Walk Test [63,<br>64] | Functional test | Baseline, follow-up | Passengers |
| Trip registration for CW | 4 | | | |
| Objective observational data from every training/trip | - Date (DD-MM-YYYY) - Duration (HH:MM) - Length (KM) - Participants (first name) - Environment of activity (e.g., park, forest, lake, urban) - Weather - Social activities (eat/drink) - Destination(s) - Mood - Overall satisfaction | Online trip registration (QR-code directing users to a short webbased questionnaire is scanned immediately after the TT or CWA- activity) | During the programme After finishing a CWA-activity. | Context related data completed by one person after each activity Passengers pilots |

# Sub-study 2. Cycling without age

Outcome and measures in the Cycling Without Age evaluation.

| Measurement (outcome) | What (operational) | How (instrument) | When (timing of collection) | Who<br>(Data source) |
|---|---|---|---|---|
| PRIMARY OUTCOME | | | | |
| Quality of life (QOL) | Cantril Ladder of Life Scale<br>[49] | Web and interview-<br>based questionnaires | Baseline, follow-up | HA, Runners,<br>Relatives |
| SECONDARY OUTCOME | S | | | |
| Autonomy | The perceived feeling of being in control over ones own life | Web-based questionnaire | Baseline, follow-up | НА |
| Sleep | Sleep quality and sleep quantity | Web-based<br>questionnaire<br>Bio tracking (HA)<br>SMS-Survey (HA) | Baseline,<br>during (HA),<br>follow-up | HA<br>Runners |
| Well-being | WHO-five Well-being<br>Index [65] | Web-based<br>questionnaire | Baseline, follow-up | HA, Runners |
| Loneliness | A perceived feeling of loneliness and lack of network and support [52, 53] | Web-based<br>questionnaire | Baseline, follow-up | HA, Runners |
| EXPLORATIVE OUTCOM | ES | I | I | |
| Self-perceived<br>health | Subjectively perceived<br>Health [54] | Web-based questionnaire | Baseline, follow-up | HA, Runners |
| Perceived pain | Mental and physical pain/discomfort [54] | Web-based<br>questionnaire | Baseline, follow-up | НА |
| Self-perceived<br>Physical performance | Subjectively perceived<br>Physical performance<br>[55] | Web-based<br>questionnaire | Baseline, follow-up | Runners |
| Epileptic seizures | Reduced epileptic seizures (adjusted version[66]) | Paper-based questionnaire | Baseline, follow-up | НА |
| Self-efficacy | General self-efficacy [56, 57] | Web-based questionnaire | Baseline, follow-up | HA, Runners |

| Measurement (outcome) | What (operational) | How (instrument) | When (timing of collection) | Who<br>(Data source) |
|---|---|---|---|---|
| Self-worth | Perceived feeling of acceptance [45] | Web-based<br>questionnaire | Baseline, follow-up | HA, Runners |
| Social/emotional support and network | Contact and support with friends, family and others. The perceived feeling of being valued, respected and accepted by others [54] | Web-based<br>questionnaire | Baseline, follow-up | НА |
| UNINTENDED SIDE EFFECT | S | | | |
| Fatigue | The perceived feeling of fatigue related to voluntariness or programme activity | Web-based<br>questionnaire | Follow-up | HA, Runners |
| Anxiety | The perceived feeling of anxiety trigged by the programme activity | Web-based<br>questionnaire | Follow-up | HA, Runners |
| Injuries | Amount of injuries by participation | Web-based<br>questionnaire | Follow-up | HA, Runners |
| Objective clinical data ( | only for HA:TT) | | | |
| Body anthropometrics | <ul> <li>Bodyweight</li> <li>Body mass index</li> <li>Whole body lean body mass</li> <li>Whole body fat mass</li> <li>Whole body bone</li> </ul> | Dual X-ray<br>absorptiometry | B1, B2 + FU | НА |
| Clinical blood samples | Blood glucose control: - HbA1c - Fasting glucose - Fasting C-peptide and insulin | Standard clinical procedure | B1, B2 + FU | НА |
| | Blood lipids: - Total cholesterol - Triglyceride | | | |
| Oral Glucose<br>Tolerance<br>Test (OGTT) | Glucose,<br>C-peptide,<br>Insulin | Standard OGTT-<br>procedure | B1, B2 + FU | НА |

| What (operational) | How (instrument) | When (timing of collection) | Who<br>(Data source) |
|---|---|---|---|
| Blood volume | Estimated from haematocrit level | B1, B2 + FU | НА |
| Resting systolic and diastolic blood pressure (pulse) | Monitored by a standard procedure for office blood pressure | B1, B2 + FU | НА |
| - Date (DD-MM-YYYY) - Duration (HH:MM) - Length (KM) - Participants (first name) - Environment of activity (e.g. park, forest, lake, urban) - Weather - Total number of participants (runners and HA) - Destination(s) | Online trip registration (QR-code directing users to a short webbased questionnaire is scanned immediately after the TT or CWAactivity) | During the programmes and after finishing a programme activity. | Context related data completed by one person after each activity TT: Runners fulfil the online form |
| | Resting systolic and diastolic blood pressure (pulse) - Date (DD-MM-YYYY) - Duration (HH:MM) - Length (KM) - Participants (first name) - Environment of activity (e.g. park, forest, lake, urban) - Weather - Total number of participants (runners and HA) | Blood volume Resting systolic and diastolic blood pressure (pulse) Date (DD-MM-YYYY) Duration (HH:MM) Length (KM) Participants (first name) Environment of activity (e.g. park, forest, lake, urban) Weather Total number of participants (runners and HA) Destination(s) Estimated from haematocrit level Monitored by a standard procedure for office blood pressure Online trip registration (QR-code directing users to a short webbased questionnaire is scanned immediately after the TT or CWA-activity) | What (operational) Blood volume Estimated from haematocrit level Resting systolic and diastolic blood pressure (pulse) Date (DD-MM-YYYY) Duration (HH:MM) Length (KM) Participants (first name) Environment of activity (e.g. park, forest, lake, urban) Weather Total number of participants (runners and HA) Destination(s) How (instrument) B1, B2 + FU B1, B2 + FU During the programmes and after finishing a programme activity. |

#### References

- 1. WHO, *World report on disability 2011*. 2011, World Health Organization: World Health Organization, 20 Avenue Appia, 1211 Geneva 27, Switzerland.
- 2. Van der Ploeg, H.P., et al., *Physical activity for people with a disability.* Sports medicine, 2004. **34**(10): p. 639-649.
- 3. Dishman, R.K., G.W. Heath, and I.-M. Lee, *Physical activity epidemiology*. 2012: Human Kinetics.
- 4. Rimmer, J.H., et al., Accessibility of health clubs for people with mobility disabilities and visual impairments. American journal of public health, 2005. **95**(11): p. 2022-2028.
- 5. Mulligan, H., M. Miyahara, and A. Nichols-Dunsmuir, *Multiple perspectives on accessibility to physical activity for people with long-term mobility impairment*. Scandinavian Journal of Disability Research, 2017. **19**(4): p. 295-306.
- 6. Ryan, J.M., et al., *The risk, burden, and management of non-communicable diseases in cerebral palsy: a scoping review.* Developmental Medicine & Child Neurology, 2018. **60**(8): p. 753-764.
- 7. Johannesen, C.K., M. Davidsen, and A.I. Christensen, Ældres sundhed og trivsel: Ældreprofilen 2019 er baseret på sundheds-og sygelighedsundersøgelserne, de nationale sundhedsprofiler og udvalgte registre. 2019: Sundhedsstyrelsen, Islands Brygge 67, 2300 København S.
- 8. Amilon, A., et al., *Personer med handicap: Hverdagsliv og levevilkår 2016*. 2017, VIVE Det Nationale Forsknings- og Analysecenter for Velfærd: Herluf Trolles Gade 11. 1052 København K.
- 9. Carroll, D.D., et al., *Vital signs: disability and physical activity—United States, 2009–2012.* MMWR. Morbidity and mortality weekly report, 2014. **63**(18): p. 407.

- 10. Whitney, D.G., et al., *Noncommunicable disease and multimorbidity in young adults with cerebral palsy*. Clinical epidemiology, 2018. **10**: p. 511.
- 11. Cremer, N., E.A. Hurvitz, and M.D. Peterson, *Multimorbidity in middle-aged adults with cerebral palsy.* The American journal of medicine, 2017. **130**(6): p. 744. e9-744. e15.
- 12. Biswas, A., et al., Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Annals of internal medicine, 2015. **162**(2): p. 123-132.
- 13. Lee, I.-M., et al., Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. The lancet, 2012. **380**(9838): p. 219-229.
- 14. Ekelund, U., et al., Does physical activity attenuate, or even eliminate, the detrimental association of sitting time with mortality? A harmonised meta-analysis of data from more than 1 million men and women. The Lancet, 2016. **388**(10051): p. 1302-1310.
- 15. Pedersen, B.K. and B. Saltin, *Exercise as medicine—evidence for prescribing exercise as therapy in 26 different chronic diseases.* Scandinavian journal of medicine & science in sports, 2015. **25**: p. 1-72.
- 16. Cunningham, C., et al., *Consequences of physical inactivity in older adults: A systematic review of reviews and meta-analyses.* Scandinavian journal of medicine & science in sports, 2020. **30**(5): p. 816-827.
- 17. Bauman, A., et al., *Updating the Evidence for Physical Activity: Summative Reviews of the Epidemiological Evidence, Prevalence, and Interventions to Promote "Active Aging"*. Gerontologist, 2016. **56 Suppl 2**: p. S268-80.
- 18. World Health Organization, *WHO guidelines on physical activity and sedentary behaviour.* 2020: Geneva.
- 19. Martin Ginis, K.A., et al., *Participation of people living with disabilities in physical activity: a global perspective.* The Lancet, 2021.
- 20. Molina-Cantero, A.J., et al., *A Study on Physical Exercise and General Mobility in People with Cerebral Palsy: Health through Costless Routines.* International Journal of Environmental Research and Public Health, 2021. **18**(17): p. 9179.
- 21. Northey, J.M., et al., *Exercise interventions for cognitive function in adults older than 50: a systematic review with meta-analysis.* British journal of sports medicine, 2018. **52**(3): p. 154-160.
- 22. Maïano, C., et al., *Exercise interventions to improve balance for young people with intellectual disabilities: a systematic review and meta-analysis*. Developmental Medicine & Child Neurology, 2019. **61**(4): p. 406-418.
- 23. Andersen, M.M., Significant experiences Development processes for young people and adults with cerebral palsy through resilience-based social adapted physical activity interventions.

  Developmental Medicine & Child Neurology, 2020. **57**: p. 1093-104.
- 24. Kissow, A.-M., *Participation in physical activity and the everyday life of people with physical disabilities: a review of the literature.* Scandinavian Journal of Disability Research, 2015. **17**(2): p. 144-166.
- 25. Kissow, A.M. and J. Singhammer, *Participation in physical activities and everyday life of people with disabilities.* European Journal of Adapted Physical Activity, 2012. **5**(2).
- 26. Ravenek, K.E., et al., Assessing quality of life in relation to physical activity participation in persons with spinal cord injury: a systematic review. Disability and health journal, 2012. **5**(4): p. 213-223.
- 27. Diaz, R., et al., *Impact of Adaptive Sports Participation on Quality of Life.* Sports Med Arthrosc Rev, 2019. **27**(2): p. 73-82.
- 28. Côté-Leclerc, F., et al., How does playing adapted sports affect quality of life of people with mobility limitations? Results from a mixed-method sequential explanatory study. Health and Quality of Life Outcomes, 2017. **15**(1): p. 22.
- 29. Vagetti, G.C., et al., Association between physical activity and quality of life in the elderly: a systematic review, 2000-2012. Brazilian Journal of Psychiatry, 2014. **36**(1): p. 76-88.

- 30. Santini, Z.I., et al., Formal social participation protects physical health through enhanced mental health: A longitudinal mediation analysis using three consecutive waves of the Survey of Health, Ageing and Retirement in Europe (SHARE). Social Science & Medicine, 2020. **251**(C).
- 31. Martin Ginis, K.A., et al., A systematic review of review articles addressing factors related to physical activity participation among children and adults with physical disabilities. Health Psychol Rev, 2016. **10**(4): p. 478-494.
- 32. Singh, M.A.F., *Exercise Comes of Age: Rationale and Recommendations for a Geriatric Exercise Prescription*. The Journals of Gerontology: Series A, 2002. **57**(5): p. M262-M282.
- 33. Rimmer, J.H., et al., Exercise intervention research on persons with disabilities: what we know and where we need to go. American Journal of Physical Medicine & Rehabilitation, 2010. **89**(3): p. 249-263.
- 34. Winther, H., et al., Forundersøgelse om Team Tvilling: Når Bevægelse Bevæger: Om betydningen af positive kropsoplevelser, ligeværdige relationer og identitetsudviklende fællesskaber for mennesker med store bevægelsesbegrænsninger. 2018, University of Copenhagen: København.
- 35. Cotnam, V., Exploring the Effects of the Cycling Without Age Program on Older Adults Living in Long-Term Care, in Health and Rehabilitation Sciences. 2020, The University of Western Ontario: Electronic Thesis and Dissertation Repository, Scholarship@Western.
- 36. Gow, A.J., C. Bell, and J. Biggar, *Cycling Without Age-Evaluation Report 2018*. 2019, Heriot Watt University UK, Dubai, Malaysia.
- 37. Gravely, E., et al., *Starting and Operating a Cycling Without Age Chapter in a Care Facility*. 2019: McMaster University, 1280 Main Street West | Hamilton, Ontario L8S4L8 | 905-525-9140.
- 38. Gray, R. and A.J. Gow, *Cycling Without Age: Assessing the Impact of a Cycling-Based Initiative on Mood and Wellbeing.* Gerontology and Geriatric Medicine, 2020. **6**: p. 2333721420946638.
- 39. McNiel, P. and J. Westphal, *Cycling without age program: the impact for residents in long-term care.* Western journal of nursing research, 2020. **42**(9): p. 728-735.
- 40. Salas, K., *Impact of "Cycling Without Age" on the health of the elderly*. 2018, HOSPITAL SANT PAUBARCELONA: Barcelona.
- 41. *Team Twin We Run Together*. 2020 [cited 2021 07/01 2021]; Available from: https://teamtvilling.dk/.
- 42. *Cycling Without Age The Right To Wind In Your Hair*. 2020 [cited 2021 18/01-2021]; Available from: <a href="https://cyklingudenalder.dk">https://cyklingudenalder.dk</a>.
- 43. *Team Tvilling [Team Twin]*. Available from: <a href="https://teamtvilling.dk">https://teamtvilling.dk</a>.
- 44. Organization, W.H., *WHOQOL*: measuring quality of life. 2019. 2019.
- 45. Jespersen, L.N., Measuring quality of life and participation in a population with diverse disabilities, in National Institute of Public Health 2018, Syddansk Universitet. Det Sundhedsvidenskabelige Fakultet: Copenhagen.
- 46. Damgaard, M., T. Steffensen, and S. Bengtsson, *Hverdagsliv og levevilkår for mennesker med funktionsnedsættelse: En analyse af sammenhængen mellem hverdagsliv, samliv, udsathed, og type og grad af funktionsnedsættelse*. 2013, VIVE: Herluf Trolles Gade 11. 1052 København K.
- 47. Levin, K.A. and C. Currie, *Reliability and validity of an adapted version of the Cantril Ladder for use with adolescent samples.* Social Indicators Research, 2014. **119**(2): p. 1047-1063.
- 48. Hinrichsen, C., et al., *Implementing Mental Health Promotion Initiatives—Process Evaluation of the ABCs of Mental Health in Denmark*. International Journal of Environmental Research and Public Health, 2020. **17**(16): p. 5819.
- 49. Cantril, H., Pattern of human concerns. 1965.
- 50. Koushede, V., et al., Measuring mental well-being in Denmark: Validation of the original and short version of the Warwick-Edinburgh mental well-being scale (WEMWBS and SWEMWBS) and cross-cultural comparison across four European settings. Psychiatry Research, 2019. **271**: p. 502-509.
- 51. Tennant, R., et al., *The Warwick-Edinburgh mental well-being scale (WEMWBS): development and UK validation.* Health and Quality of life Outcomes, 2007. **5**(1): p. 63.

- 52. Russell, D., L.A. Peplau, and C.E. Cutrona, *The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence.* Journal of personality and social psychology, 1980. **39**(3): p. 472.
- Hughes, M.E., et al., A short scale for measuring loneliness in large surveys: Results from two population-based studies. Research on aging, 2004. **26**(6): p. 655-672.
- 54. Jensen, H.A.R., et al., *Danskernes sundhed-Den nationale sundhedsprofil 2017*. 2018, National Institute of Public Health: Islands Brygge 67, 2300 København S
- 55. Grimby, G., et al., *The "Saltin–Grimby physical activity level scale" and its application to health research.* Scandinavian journal of medicine & science in sports, 2015. **25**: p. 119-125.
- 56. Schwarzer, R. and M. Jerusalem, *Generalized self-efficacy scale*. Measures in health psychology: A user's portfolio. Causal and control beliefs, 1995. **1**(1): p. 35-37.
- 57. Nielsen, L., et al., *Måling af mental sundhed: En baggrundsrapport for spørgeskemaundersøgelsen Danskernes Trivsel 2016*. 2017, University of Southern Denmark Øster Farimagsgade 5A, 2. sal, 1353 København K.
- 58. Jørgensen, K., et al., *Brief Assessment of Impaired Cognition Questionnaire (BASIC-Q)—*Development and validation of a new tool for identification of cognitive impairment in community settings. International journal of geriatric psychiatry, 2020. **35**(7): p. 693-701.
- 59. Jørgensen, K., et al., Validation of the Brief Assessment of Impaired Cognition and the Brief Assessment of Impaired Cognition Questionnaire for identification of mild cognitive impairment in a memory clinic setting. International journal of geriatric psychiatry, 2020. **35**(8): p. 907-915.
- 60. Guralnik, J.M., et al., Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. The Journals of Gerontology Series A: Biological Sciences and Medical Sciences, 2000. **55**(4): p. M221-M231.
- 61. *Short Physical Performance Battery (SPPB)*. [cited 2021 21/6 2021]; Available from: https://www.nia.nih.gov/research/labs/leps/short-physical-performance-battery-sppb.
- 62. Suetta, C., et al., *The Copenhagen Sarcopenia Study: lean mass, strength, power, and physical function in a Danish cohort aged 20–93 years.* Journal of cachexia, sarcopenia and muscle, 2019. **10**(6): p. 1316-1329.
- 63. Laboratories, A.C.o.P.S.f.C.P.F., *ATS statement: guidelines for the six-minute walk test.* Am J Respir Crit Care Med, 2002. **166**: p. 111-117.
- 64. Du, H., et al., A review of the six-minute walk test: its implication as a self-administered assessment tool. European journal of cardiovascular nursing, 2009. **8**(1): p. 2-8.
- 65. Bech, P., Subjective positive well-being. World Psychiatry, 2012. **11**(2): p. 105.
- 66. Midtjylland, N.A.-R. *SPØRGESKEMA OM DIN EPILEPSI* 2011 [cited 2021 15/07-2021]; Available from: <a href="https://docplayer.dk/16414548-Spoergeskema-om-din-epilepsi.html">https://docplayer.dk/16414548-Spoergeskema-om-din-epilepsi.html</a>.